CLINICAL TRIAL: NCT02481349
Title: Couple-Based Yoga Program for Glioma Patients and Their Partners
Brief Title: Couples-Based Yoga Program in Improving Quality of Life in Patients With High-Grade Glioma Undergoing Radiation Therapy and Their Partners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0013; NCI-2015-01124 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0013 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Caregiver; Glioma
MeSH Terms: conditions — Glioma | interventions — Practice Guidelines as Topic; Standard of Care; Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (couple-based Hatha yoga program) (Experimental): Patients and their partners attend up to 15, 45-60 minute sessions of Hatha yoga over the course of radiation therapy 5 times a week for 5-6 weeks. The program comprises four main components: joint loosening with breath synchronization; postures with deep relaxation techniques; breath energization with sound resonance; and meditation. At the fifth session, patients and their partners receive a DVD and are encouraged to practice on their own (individually and/or together) on the days when they do not meet with the instructor.
  Interventions: Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Yoga
- Arm II (waitlist control) (Active Comparator): Patients receive standard of care provided by the health care team and complete questionnaires before and after radiation therapy.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II (waitlist control)
Other: Informational Intervention — Receive DVD for home practice
  Arms: Arm I (couple-based Hatha yoga program)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Yoga — Complete couple-based Hatha yoga program
  Other Names: Yoga Therapy
  Arms: Arm I (couple-based Hatha yoga program)

SUMMARY:
This randomized clinical trial studies couples-based yoga program in improving quality of life in patients with high-grade glioma undergoing radiation therapy and their partners. A couple-based Hatha yoga program may improve fatigue, distress, sleep quality, and overall quality of life in patients with glioma and their partners.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine the feasibility of a couple-based and a caregiver yoga program in glioma patients undergoing radiotherapy (RT) and their partners.

SECONDARY OBJECTIVES:

I. Establish the initial efficacy of the yoga program in patients and their partners regarding quality of life (QOL) outcomes (i.e., fatigue, sleep disturbance, depressive symptoms, and overall QOL and health care utilization).

EXPLORATORY OBJECTIVES:

I. Explore potential moderation (e.g., baseline psychological distress, patients' tumor grade, performance status and class attendance) of the intervention effects.

OUTLINE: The first five couples are assigned to arm I. All subsequent couples are randomized to 1 of 2 arms.

ARM I: Patients and their partners attend up to 15, 45-60 minute sessions of Hatha yoga over the course of radiation therapy 5 times a week for 5-6 weeks. The program comprises four main components: joint loosening with breath synchronization; postures with deep relaxation techniques; breath energization with sound resonance; and meditation. At the fifth session, patients and their partners receive a digital video disc (DVD) and are encouraged to practice on their own (individually and/or together) on the days when they do not meet with the instructor.

ARM II: Patients receive standard of care provided by the health care team and complete questionnaires before and after radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and speak English
* Able to provide informed consent
* PATIENTS ONLY: Diagnosed with a primary glioma and going to receive at least 4 weeks of radiotherapy with at least 20 fractions
* PATIENTS ONLY: Karnofsky performance status (KPS) of 80 or above
* PATIENTS ONLY: Having an informal caregiver (spouse, romantic partner, adult child, sibling, or friend) who is willing to participate; for phase 1 only, if patients do not have one consistent primary caregiver for the duration of the study, they may be accompanied to the yoga sessions by an alternate caregiver who meets eligibility criteria

Exclusion Criteria:

* PATIENTS ONLY: for phase 1 only, regularly (self-defined) participated in a yoga practice in the year prior to diagnosis
* PATIENTS ONLY: for phase 1 only, physician-rated life expectancy of less than 6 months
* PATIENTS ONLY: for phase 1 and 2, cognitive deficits that would impede the completion of self-report instruments as deemed by the clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a couple-based yoga program, determined by overall accrual | Up to 6 weeks
Feasibility of a couple-based yoga program, determined by attrition using the Mental Component Summary of Short Form-36 | Up to 6 weeks
  The questionnaires ask about health, any symptoms, mood, level of fatigue, sleeping habits, relationship, and quality of life.
  Scale answers range from: All of the time, Most of the time, Some of the time, A little of the time, None of the time.
Feasibility of a couple-based yoga program determined by adherence | Up to 6 weeks
  Trial determined feasible if 1) ≥ 50% of eligible couples consent (i.e., approach 80 couples to obtain 40 consents in phase 1 and approach 150 dyads to achieve 75 that consent in phase 2); 2) ≥ 70% of enrolled couples complete all assessments; 3) on average ≥ 50% of all practice sessions are attended; 4) no attributable AE or SAE occur
Feasibility of a couple-based yoga program, determined by incidence of adverse events and serious adverse events | Up to 6 weeks

SECONDARY OUTCOMES:
Preliminary evidence of intervention efficacy, measured by answers on change in quality of life (QOL): SF-36 questionnaire | Up to 6 weeks
  Question answers range : All of the time, Most of the time, Some of the time, A little of the time, None of the time

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, MA,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Snyder S, Silva RF, Whisenant MS, Milbury K. Videoconferenced Yoga Interventions for Cancer Patients and their Caregivers during the COVID-19 Pandemic: A Report from a Clinician's Perspective. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211019111. doi: 10.1177/15347354211019111. PMID 34036820
- [Derived] Milbury K, Li J, Weathers SP, Mallaiah S, Armstrong T, Li Y, Bruera E, Cohen L. Pilot randomized, controlled trial of a dyadic yoga program for glioma patients undergoing radiotherapy and their family caregivers. Neurooncol Pract. 2019 Jul;6(4):311-320. doi: 10.1093/nop/npy052. Epub 2018 Dec 20. PMID 31386042
- [Derived] Milbury K, Li J, Weathers SP, Shih T, Malliaha S, Li Y, Cohen L. A research protocol for a pilot, randomized controlled trial designed to examine the feasibility of a dyadic versus individual yoga program for family caregivers of glioma patients undergoing radiotherapy. Pilot Feasibility Stud. 2019 Jul 25;5:95. doi: 10.1186/s40814-019-0479-5. eCollection 2019. PMID 31367462
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org